CLINICAL TRIAL: NCT03457350
Title: Small-caliber Office Hysteroscopy Versus Blind Cervical Probing for Tight Primary Cervical Stenosis in Nulliparous Women: a Preliminary Study
Brief Title: Office Hysteroscopy Versus Cervical Probing for Cervical Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor Dr Atef Darwish MD PhD, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: hysteroscopy versus probing
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Hysteroscopy
Keywords: hysteroscopy; cervical stenosis; probing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- office hysteroscopy (Experimental): Office hysteroscopy 30 degrees 2.6 mm telescope with an outer sheath of 3.2 mm (Storz Co., Tutlingen, Germany). Hysteroscopy is performed as usual by proper examination of the vagina and the ectocervix for any abnormality followed by introduction of the hysteroscope into the cervical canal. At this step, the hysteroscopist waits for a while until the distending fluid forms a micro-cavity. At this point, the telescope is advanced with necessary rotatory movements of the 30 degrees telescope guided by the vision of the dark spot which is the internal os. If it is reached, again waiting for some time to allow fluid distension of the internal os area.
  Interventions: Procedure: cervical negotiation
- blind cervical probing (Experimental): Cervical probing is started with a 2 mm probe after grasping the cervix with a multi-tooth tenaculum put anteriorly or posteriorly according to prior transabdominal or transvaginal sonographic examination of the cervical canal. If the probe succeedes to bypass the internal os, a higher caliber probe is used. Thereafter, a uterine sound (4mm = 1.33 Fr) is introduced into the endometrial cavity. Lastly, gentle cervical dilatation up to Hegar's 8 is performed as usual with classic leaving each dilator for 30 seconds inside the internal os. If probes couldn't bypass the internal os, the procedure is considered failed. If the probe enters a cavity other than endometrial cavity, a false passage is considered.
  Interventions: Procedure: cervical negotiation

INTERVENTIONS:
Procedure: cervical negotiation — trial to bypass severe cervical stenosis

SUMMARY:
This study aims to estimate if performing a small caliber office hysteroscopic cervical negotiation would succeed to bypass tight markedly stenotic cervix in comparison to blind cervical probing done under general anesthesia. Moreover, the investigators test the impact of drawing a detailed diagram after this procedure on the success of ET in participants with failed mock or actual trials of embryo transfer (ET).

DETAILED DESCRIPTION:
It comprises 122 nulliprous women with failed cervical sounding on vaginal examination in the office. Participants were divided into 2 groups. Group A comprised 64 cases subjected to small-caliber office hysteroscopic cervical negotiation while 58 cases were subjected to cervical probing under general anesthesia. Main outcome measures included success to bypass primary cervical stenosis and complication rate

ELIGIBILITY:
Inclusion Criteria:

* Nulliprous women.
* Failed cervical sounding on vaginal examination in the office.

Exclusion Criteria:

* Previous operation on the cervix.
* Use of any medication to prime the cervix (primary).
* Multiparity: weather delivered vaginally or by cesarean sectrion

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
How many cases of access to the endometrial cavity | 20 minutes
  overcoming cervical stenosis

SECONDARY OUTCOMES:
complication rate | 20 minutes
  how many cases with perforation or false passage

CONTACTS AND LOCATIONS:
Overall Officials: Atef Darwish, Principal Investigator — Woman's |Health University Hospital
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No